CLINICAL TRIAL: NCT05297097
Title: The Impact of a Human Breast Milk Supplement on Epigenetic and Cellular Markers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TruDiagnostic (Industry)
Collaborators: Adventa Biosciences (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AB-BMA-001
Record Dates: First submitted 2022-03-10; First posted 2022-03-28 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: single arm, prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trulacta breastmilk supplement (Experimental): Once daily Trulacta supplement
  Interventions: Dietary Supplement: Trulacta breastmilk supplement

INTERVENTIONS:
Dietary Supplement: Trulacta breastmilk supplement — one supplement daily

SUMMARY:
This is a trial to assess the effects of the Trulacta supplement on biological age, sleep quality, immune system and wellness markers.

DETAILED DESCRIPTION:
Human breast milk has been widely studied in babies, as have certain elements of breast milk in adults. None of those studies, however, address the effectiveness of raw breast milk in adults. Furthermore, Adventa Bioscience's proprietary process of converting breast milk into a powder which is then encapsulated has not been studied. Early customers of the breast milk capsule, Trulacta, have experienced incredible results; from increased sleep, reduced pain and bloating, and reduction or elimination of symptoms caused by severe diseases. An early analysis of Trulacta in partnership with a company 4Life, has shown that the milk powder in Trulacta has a high immunologic activity level with Natural Killer cells in controlled environment.

The purpose of this non-randomized, prospective clinical trial is to evaluate the effect of 90 days of supplementation with a human breast milk supplement on sleep quality, low-grade chronic inflammation, immuno-modulation, metabolic health, and epigenetic aging.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of any ethnicity.
* Age Range - 18 - 85 years (inclusive)
* Participant must be able to comply with treatment plan and laboratory tests
* Participant must be able to read, write, and speak English fluently
* Participant must have an established primary care provider
* Participant must be willing and able to consume 2 capsules per day throughout the duration of study period
* Participant must have a mobile telephone and internet connection

Exclusion Criteria:

* Patients with a self-reported history of lactose intolerance
* History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Known immune system issues or immunodeficiency disease
* History of viral illness which could be reactivated by immune downregulation
* Presence of clinically significant acute or unstable cardiovascular and cerebrovascular (stroke) disease
* Diagnosis of a transient ischemic attack in the 6 months prior to screening
* Participants infected with hepatitis C or HIV
* Presence of active infection in previous 4 weeks
* Any other illness, psychiatric disorder, alcohol or chemical dependence that in the opinion of the Clinical Investigator would render a participant unsuitable to participate in the study
* Unable or unwilling to provide required blood sample for testing
* Current or previous use of known prescription immunomodulating products (e.g. glucocorticoids, TNF-alpha inhibitors) in the month prior to the start of the trial.
* A known history of blood dyscrasias including coagulopathy
* Current pregnancy, planned attempts to conceive during study period or sexually active females not using contraception, as well as lactating/nursing females
* Any person deemed by Clinical Investigator as low likelihood of complying with study protocol (e.g. evidence of history of non-compliance, history of poor follow-up, multiple or complex scheduling conflicts).
* Planned surgical procedure during study period
* Participants who are actively engaged in weight-loss or have started any new medications during the duration of the trial that can potentially interfere with the study, as deemed appropriate by Primary Clinical Investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Epigenetic Age | Testing will compare results from baseline to completion of 3 months of the supplement
  DNA methylation testing completed with 850kEPIC array

SECONDARY OUTCOMES:
Sleep Quality | Assessment will compare baseline with testing completed after 3 months of the supplement
  Patients will complete the Pittsburgh Sleep Quality Index (PSQI) at baseline, monthly, and after completing the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Central Florida Wellness, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Esser N, Legrand-Poels S, Piette J, Scheen AJ, Paquot N. Inflammation as a link between obesity, metabolic syndrome and type 2 diabetes. Diabetes Res Clin Pract. 2014 Aug;105(2):141-50. doi: 10.1016/j.diabres.2014.04.006. Epub 2014 Apr 13. PMID 24798950
- [Background] Oudi ME, Aouni Z, Mazigh C, Khochkar R, Gazoueni E, Haouela H, Machghoul S. Homocysteine and markers of inflammation in acute coronary syndrome. Exp Clin Cardiol. 2010 Summer;15(2):e25-8. PMID 20631860